CLINICAL TRIAL: NCT04141436
Title: Open Label, Randomized Controlled Trial, Effect of Hypnofertility on Fertility Preparedness, Cortisol Levels and Pregnancy Outcomes of Women Undergoing In Vitro Fertilization
Brief Title: Hypnofertility for Women Undergoing In Vitro Fertilization (HWUIVF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sevcan Fata, Director, Clinical research, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DOKUZ12345
Record Dates: First submitted 2019-10-10; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Infertility Unexplained; Fertility Disorders
Keywords: Hypnofertility; fertility preparedness; cortisol level; pregnancy outcome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention Based on Hypnofertility
  Interventions: Behavioral: Interventions Based on Hypnofertility
- Control (Active Comparator): Routine clinical procedure
  Interventions: Other: Routine clinical procedure

INTERVENTIONS:
Behavioral: Interventions Based on Hypnofertility — Affirmation Visualization Imagination Relaxation
  Arms: Intervention
Other: Routine clinical procedure — Routine clinical procedure
  Arms: Control

SUMMARY:
This randomized controlled study aimed to specify whether the interventions based on Hypnofertility would lead to increased fertility preparedness and pregnancy outcomes, decreased cortisol levels of women undergoing In Vitro Fertilization (IVF) treatment.

DETAILED DESCRIPTION:
Objective: To specify whether the interventions based on Hypnofertility would lead to increased fertility preparedness and pregnancy outcomes, decreased cortisol levels of women undergoing In Vitro Fertilization (IVF) treatment.

Design: Randomized, controlled, prospective study. Setting: University Hospital Fertility Center in Izmir. Patients: Sixty-one women with unexplained infertility undergoing IVF treatment.

Interventions: Interventions based on Hypnofertility including affirmations, visualization, dreaming and relaxation from the first day of treatment to the day of pregnancy test.

Main Outcome Measures: Fertility preparedness and cortisol levels (primary outcomes), pregnancy rate (secondary outcome).

ELIGIBILITY:
Inclusion Criteria:

* primary infertility,
* unexplained infertility,
* going to undergo IVF treatment,
* fresh embryos,
* under 39 years of age
* having a smart phone

Exclusion Criteria:

* participated in any program to reduce stress
* having any psychiatric disorder

Max Age: 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Fertility preparedness | through study completion, average 28 days
  Fertility Preparedness Scale for Women Receiving Fertility Support (FPS) The 5-point Likert scale was developed by Fata and Aluş Tokat (Fata and Aluş Tokat, 2019). This scale items consist only of positive words. The scale consists of 3 sub-dimensions: "Hope and Awareness"," Positive Feelings and Thoughts ","Prepared Body and Brain". Since the items consisted only of positive expressions, the score was calculated as they were. The scores of the items were 5 (strongly agree), 4 (agree), 3 (neutral), 2 (disagree) and 1 (strongly disagree), respectively. The minimum and maximum scores are 23 and 115, respectively. The median of the scale score is 56 points, which can be considered the cut value. If the scale score is below 56, it can be considered that the woman is not prepared for fertility. If the score is 56 and higher, it indicates greater fertility preparedness.
cortisol levels | through study completion, average 28 days
  The saliva samples were collected in sterile urine containers provided by the researcher and stored in the refrigerator at a temperature between +4 and +8 degrees for a maximum of two (2) months. On average, they were sent to the laboratory every 15 days by means of carrying bags containing ice molds. Saliva was studied by LC-MS/MS (Liquid Chromatography-Mass Spectrometry) method by the expert staff of the laboratory.
  Cortisol level (nmol/L) measurement was obtained for both intervention and control group in all face-to-face sessions. Because cortisol level have diurnal rythm and highest level is shown in the morning, samples were of all women in the morning once they came to clinic. Samples were to be collected with no eating, drinking, gum chewing or smoking in the 30 minutes prior to collection.

SECONDARY OUTCOMES:
pregnancy rate | through study completion, average 28 days
  result of pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Sevcan Fata, Principal Investigator — Dr.
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)